CLINICAL TRIAL: NCT04292171
Title: Gabapentin for Perioperative Pain Relief in Surgical Abortion: a Double-blind Randomized Controlled Trial
Brief Title: Gabapentin for Perioperative Pain Relief in Surgical Abortion
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Nevada, Las Vegas (Other)
Responsible Party: Principal Investigator, Adam Levy, Associate Professor, OB/GYN, University of Nevada, Las Vegas
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 734275-7
Record Dates: First submitted 2020-02-05; First posted 2020-03-02 (Actual); Results first posted 2020-12-02 (Actual); Last update posted 2020-12-02 (Actual); Status verified 2020-11

CONDITIONS: Pain Control
Keywords: Gabapentin Abortion
MeSH Terms: conditions — Agnosia | interventions — Gabapentin

STUDY DESIGN:
Intervention Model Description: double-blind placebo-controlled randomized controlled trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: pharmacy prepared sequentially numbered opaque bottles with identical capsules containing either placebo (vit c) or Gabapentin 600mg, block randomized
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Gabapentin Arm (Active Comparator): Gabapentin 600 mg given 1-2 hours prior to surgical abortion
  Interventions: Drug: Gabapentin
- Placebo Arm (Placebo Comparator): Placebo (vit C) given 1-2 hours prior to surgical abortion
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Gabapentin — Preoperative treatment with Gabapentin
  Arms: Gabapentin Arm
Drug: Placebos — Preoperative treatment with Placebo
  Arms: Placebo Arm

SUMMARY:
Gabapentin preoperative use for evaluation of benefit to reduce pain during and after surgical office-based abortion.

DETAILED DESCRIPTION:
A double-blind placebo controlled trial of gabapentin in the setting of an ambulatory surgical abortion center where patients receive either the routine intravenous sedation, local cervical anesthesia plus 600mg of gabapentin one hour prior to surgery vs. the same regimen plus placebo one hour prior to surgery. Our primary outcome measure will be post-operative validated pain scores using a 11-point visual analog scale (VAS). Secondary measures will include nausea and vomiting during, after and 24 hours after the procedure. A second and third pain assessment using VAS will be made at 30 minutes and at 24 hours postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Women seeking surgical abortion between 5 and 23 6/7 weeks of ultrasound age.
* English or Spanish speaking
* eligible for office-based surgical pregnancy termination

Exclusion Criteria:

* present use of gabapentin or pregabalin,
* renal disease
* sensitivity or allergy to gabapentin
* Missed abortion

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 219 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2018-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vani Dandolu, MD, Study Chair — University of Nevada School of Medicine
Locations (1):
- Birth Control Care Center, Las Vegas, Nevada, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the participant data de-identified that was collected during the study.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Following publication and terminating 5 years following
Access Criteria: Investigators must submit a Material Transfer Agreement for data transfer between UNLV School of Medicine and investigators institution. Investigators who demonstrate a legitimate proposal on the purpose for the data set, their intended analysis and schedule for anticipated publication will be considered. Investigators should submit their publications within 18 months of receiving the data set.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Gabapentin Arm | Placebo Arm
Started | 109 | 110
Completed | 107 | 109
Not Completed | 2 | 1
Not completed — Pharmacy error | 2 | 0
Not completed — Delivered prior to procedure | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gabapentin Arm | Placebo Arm | Total
Number analyzed (Participants) | 107 | 109 | 216
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.7 (6.26) | 27.1 (6.03) | 27.4 (6.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 107 | 109 | 216
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic/Latino | 36 | 47 | 83
  White/Caucasian | 53 | 39 | 92
  Black/ African American | 20 | 18 | 38
  Asian | 6 | 5 | 11
  Hawiian/Pacific Islander | 3 | 0 | 3
  other | 17 | 33 | 50
  more than one | 3 | 10 | 13
Region of Enrollment [Number; unit: participants]
  United States | 107 | 109 | 216
Pregnancy History [Count of Participants; unit: Participants]
  Previous Pregnancy "YES" | 82 | 88 | 170
  History of Vaginal deliveries | 40 | 59 | 99
  History of cesarean delivery | 18 | 23 | 41
  History of Abortions | 51 | 47 | 98
  History of Miscarriages | 23 | 20 | 43
  History of Stillbirths | 0 | 4 | 4
  history of ectopic pregnancy | 0 | 5 | 5
  History of Surgical Abortion | 46 | 44 | 90
Living Arrangements [Count of Participants; unit: Participants]
  Alone | 13 | 10 | 23
  with Partner | 44 | 46 | 90
  with Children | 28 | 44 | 72
  with Friends | 7 | 7 | 14
  with Family | 37 | 35 | 72

OUTCOME MEASURES:

1. Primary Outcome: Pain Score
Description: 100mm Visual analog scale (VAS) for level of pain, 1-100, 1=no pain, 100= extreme pain
Time Frame: 5 minutes postoperative
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Gabapentin Arm | Placebo Arm
Number analyzed (Participants) | 107 | 109
score on a scale | 17 [0 to 60] | 17 [2 to 53]

2. Secondary Outcome: Pain Score 24
Description: Pain at 24 hours postoperative on 100mm VAS, 1=no pain, 100=extreme pain
Time Frame: 24 hours postop
Population: We lost to followup 40 in Gaba arm, 48 in the placebo arm at 24 hrs - these patients did not respond to our calls
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Gabapentin Arm | Placebo Arm
Number analyzed (Participants) | 67 | 61
score on a scale | 0 [0 to 20] | 1 [0 to 12.5]

3. Secondary Outcome: Nausea
Description: Nausea at 24 hours using 100mm VAS, 1=none, 100=extreme
Time Frame: 24 hours postoperative
Measure: Mean (Standard Deviation); unit: VAS 100mm
Arm/Group | Gabapentin Arm | Placebo Arm
Number analyzed (Participants) | 68 | 61
VAS 100mm | 1.74 (10.923) | 1.74 (8.140)

4. Secondary Outcome: Vomiting
Description: Vomiting at 24 hrs, 100mm VAS, 1=none, 100=extreme
Time Frame: 24 hours postoperative
Measure: Mean (Standard Deviation); unit: VAS 100mm
Arm/Group | Gabapentin Arm | Placebo Arm
Number analyzed (Participants) | 68 | 61
VAS 100mm | 0.85 (6.063) | 0.74 (5.125)

5. Secondary Outcome: Pain Score at 30 Minutes Postoperative
Description: 100mm Visual analog scale for level of pain, 1-100, 1=no pain, 100= extreme pain
Time Frame: 30 minutes postoperative
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Gabapentin Arm | Placebo Arm
Number analyzed (Participants) | 107 | 109
score on a scale | 20 [3 to 55] | 23 [3 to 57]

ADVERSE EVENTS:
Time Frame: 24 hours
Description: There were no reported adverse event in the study groups
Arm/Group | Gabapentin Arm | Placebo Arm
All-Cause Mortality (participants affected / at risk) | 0/107 | 0/109
Serious Adverse Events (participants affected / at risk) | 0/107 | 0/109
Other Adverse Events (participants affected / at risk) | 0/107 | 0/109

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-01): https://cdn.clinicaltrials.gov/large-docs/71/NCT04292171/Prot_SAP_000.pdf